CLINICAL TRIAL: NCT05007977
Title: Pharmacodynamic Evaluation of ZT-01 in a Stepped Hypoglycemic Clamp Model in Subjects With Type 1 Diabetes Mellitus
Brief Title: Effect of ZT-01 on Glucagon During Hypoglycemia in Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was completed following review of the assumptions underlying the power calculation and it was deemed that enough subjects had been recruited to complete enrollment
Sponsor: Zucara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZT01-CL-1003
Record Dates: First submitted 2021-07-20; First posted 2021-08-17 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: hypoglycemic clamp; glucagon counterregulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to the order in which they receive three treatments during consecutive clamps
Who Masked: Participant, Investigator
Masking Description: The participant, the investigator and site staff conducting all study procedures are masked to treatment administered at each clamp.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment order: placebo, low dose, high dose (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo
- Treatment order: placebo, high dose, low dose (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo
- Treatment order: low dose, placebo, high dose (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo
- Treatment order: low dose, high dose, placebo (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo
- Treatment order: high dose, placebo, low dose (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo
- Treatment order: high dose, low dose, placebo (Experimental): Subjects will receive a single administration of each treatment in this order during three consecutive clamps
  Interventions: Drug: ZT-01 low dose; Drug: ZT-01 high dose; Drug: Placebo

INTERVENTIONS:
Drug: ZT-01 low dose — Single subcutaneous (SC) injection of ZT-01 3 mg during hypoglycemic clamp
Drug: ZT-01 high dose — Single SC injection of ZT-01 20 mg during hypoglycemic clamp
Drug: Placebo — Single SC injection of placebo during hypoglycemic clamp

SUMMARY:
The purpose of this study is to determine whether ZT-01 increases the glucagon response to hypoglycemia in type 1 diabetes (T1D). ZT-01 is a specific somatostatin (SST) type 2 receptor antagonist hypothesized to increase the counterregulatory glucagon release during hypoglycemia, which is impaired in diabetes, and may thus reduce the occurrence of hypoglycemia.

Approximately 25 participants with well-controlled type 1 diabetes will be recruited to a crossover study and be randomized to the order in which they receive a single administration of placebo, low dose and high dose ZT-01 during three euglycemic-hypoglycemic clamps 2 to 6 weeks apart, with a follow-up visit approximately 1 week after the final clamp.

Participants will stay overnight in the clinic before each clamp, and their plasma glucose (PG) will be kept at euglycemic levels with IV insulin and dextrose as needed. The following morning, the clamp will begin and the subject's PG will be kept at 5.5 mmol/L (euglycemia) with variable IV insulin (and dextrose as needed). Study treatment will be administered during this euglycemic period, and then insulin will be increased so that PG falls to a plateau of mild hypoglycemia, and then increased further to clinically significant hypoglycemia. Release of glucagon and other counterregulatory hormones will be measured, and a symptom score will be completed, during euglycemia before and following study treatment, and during each level of hypoglycemia. Following the clamp, the participant's blood glucose will be returned to normal levels prior to leaving the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 5 years and receiving insulin as the only T1D therapy
* HbA1c ≥6.0 and ≤9.0 %
* BMI ≥18 to ≤27 kg/m^2
* Normal thyroid function

Exclusion Criteria:

* Impaired hypoglycemia awareness
* Severe hypoglycemia or diabetic ketoacidosis (DKA) within 3 months
* Abnormal blood pressure or ECG, clinically significant cardiovascular, cerebrovascular or peripheral vascular disease
* History of pheochromocytoma, insulinoma, glucagonoma, acromegaly, Cushing's disease, glycogen storage disease or adrenal insufficiency; ongoing or previous treatment with octreotide, lanreotide or pasireotide
* Current use of systemic corticosteroids or beta-blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Change in glucagon between euglycemia and hypoglycemia | During each clamp, up to 12 weeks
  Mean and peak glucagon level during euglycemia and each hypoglycemic period of the clamp

SECONDARY OUTCOMES:
Insulin infused | During each clamp, up to 12 weeks
  Insulin administered during euglycemia and each hypoglycemic period of the clamp
Insulin infusion rate | During each clamp, up to 12 weeks
  Rate of insulin administered during euglycemia and each hypoglycemic period of the clamp
Change in catecholamines between euglycemia and hypoglycemia | During each clamp, up to 12 weeks
  Epinephrine and norepinephrine during euglycemia and each stable hypoglycemic period of the clamp
Change in growth hormone between euglycemia and hypoglycemia | During each clamp, up to 12 weeks
  Growth hormone during euglycemia and each stable hypoglycemic period
Change in cortisol between euglycemia and hypoglycemia | During each clamp, up to 12 weeks
  Cortisol during euglycemia and each stable hypoglycemic period

OTHER OUTCOMES:
Symptom score during hypoglycemia | During each clamp, up to 12 weeks
  The Edinburgh hypoglycemia symptom score assesses the presence and extent (on a scale of 1, not present to 7, present a great deal) of 16 common symptoms which may be experienced by an individual while their blood glucose is low. The score does not indicate any outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Liggins, PhD, Study Director — Zucara Therapeutics Inc.
Locations (1):
- LMC Manna Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No